CLINICAL TRIAL: NCT01977352
Title: Comparison of Cumulative Opioid Consumption After Interscalene Brachial Plexus Block With Liposomal Bupivacaine (Exparel; 88 mg in 20 cc) Versus Bupivacaine 0.25% for Arthroscopic Shoulder Surgery
Brief Title: Efficacy of Interscalene Brachial Plexus Block With Liposomal Bupivacaine for Arthroscopic Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-0064
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Shoulder Pain; Rotator Cuff Tear
Keywords: Exparel; Liposomal Bupivacaine; Arthroscopic Shoulder Surgery
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine 0.25% (Active Comparator): 20 cc of bupivacaine 0.25%
  Interventions: Drug: Liposomal bupivacaine
- Liposomal bupivacaine (Experimental): liposomal bupivacaine (EXPAREL®; 88 mg in 20 cc)
  Interventions: Drug: Bupivacaine 0.25%

INTERVENTIONS:
Drug: Liposomal bupivacaine — liposomal bupivacaine (EXPAREL®; 88 mg in 20 cc)
  Other Names: Exparel
  Arms: Bupivacaine 0.25%
Drug: Bupivacaine 0.25% — 20 cc of bupivacaine 0.25%
  Other Names: Bupivacaine
  Arms: Liposomal bupivacaine

SUMMARY:
The purpose of this study is to compare the quality and duration of pain relief after shoulder surgery provided by a single injection of liposomal bupivacaine versus standard bupivacaine when administered as an interscalene brachial plexus block. It is hypothesized that the liposomal bupivacaine formulation will provide more effective pain relief than standard bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults (age >17 years) of American Society of Anesthesiologists (ASA) I-III physical class scheduled for elective arthroscopic shoulder surgery will be eligible to participate regardless of race/ethnicity.

Exclusion Criteria:

* Subjects will not be eligible for this trial if they report a history of an allergy to a local anesthetic, baseline neurological deficit, a medical condition that would make it difficult to assess sensory distribution or communicate with the staff, a recent history (< 3 months) of drug or alcohol abuse, concomitant opioid therapy, or a preexisting coagulation disorder.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shariat, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's Roosevelt Hospital Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Bupivacaine 0.25%
Started | 21 | 21
Completed | 20 | 19
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Bupivacaine 0.25% | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (9.55) | 54.69 (9.45) | 55.1 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption
Description: Compare total opioid consumption up to 1 week post operatively between patients receiving bupivacaine 0.25% (20 cc) and liposomal bupivacaine (EXPAREL®; 88 mg in 20 cc) for interscalene brachial plexus block.
Time Frame: Post op Day 1, post op Day 2, post op day 3, post op 1 week
Measure: Mean (Standard Deviation); unit: number of percocet tabs
Arm/Group | Liposomal Bupivacaine | Bupivacaine 0.25%
Number analyzed (Participants) | 20 | 19
number of percocet tabs
  Post op Day 1 | 2 (1.53) | 2.75 (2.96)
  Post op Day 2 | 1.94 (1.47) | 3.33 (3.61)
  Post op Day 3 | 2.06 (2.01) | 3.63 (3.7)
  Post Op 1 Week | 1.61 (1.61) | 1.13 (2.03)

2. Secondary Outcome: Quality of Analgesia
Description: The Numeric Rating Scale (NRS-11) is an 11-point scale, from 0 = no pain to 10 = Severe Pain, for patient self-reporting of pain.
Time Frame: Post op Day 1, post op Day 2, post op day 3, post op 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine 0.25%
Number analyzed (Participants) | 20 | 19
units on a scale
  Post op Day 1 | 5.23 (3.5) | 6.4 (2.15)
  Post op Day 2 | 4.9 (3.4) | 6.13 (2.66)
  Post op Day 3 | 5.18 (2.77) | 5.14 (3.08)
  Post Op 1 Week | 4.08 (2.88) | 3.66 (2.46)

3. Secondary Outcome: Sensory and Motor Block
Description: Measurement of brachial plexus blockade upon completion of the peripheral nerve block and prior to surgery. Sensory block will be assessed by pinprick with a paper clip using a 1-3 scale: 1, no block (complete sensation); 2, parasthesia (light touch); 3, anesthesia (no sensation). Motor block uses the same 1-3 scale: 1 = no block, 2= parasthesia and 3=anesthesia. Evaluation of sensory block will also be undertaken at one after arrival to the Post Anesthesia Care Unit (PACU). The first occurrence of pain perceived by the patient will be used as a surrogate for return of the sensory function.
Time Frame: at 20 min and at 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine 0.25%
Number analyzed (Participants) | 20 | 19
units on a scale
  Sensory block at 20 min prior to surgery | 1.6 (0.43) | 1.31 (0.42)
  Motor block at 20 min prior to surgery | 2.8 (0.43) | 2.33 (0.7)
  Sensory block at 1 hour after arrival to PACU | 1.78 (2.77) | 1.08 (2.08)

4. Secondary Outcome: Time to First Pain Medicine
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Liposomal Bupivacaine | Bupivacaine 0.25%
Number analyzed (Participants) | 20 | 19
minutes | 1148 (1227.59) | 702.89 (273.06)

5. Secondary Outcome: Time to Discharge Home
Description: data not collected
Time Frame: 72 hours
Arm/Group | Liposomal Bupivacaine | Bupivacaine 0.25%
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Incidence of Postoperative Nausea and Vomiting
Time Frame: 72 hours
Measure: Number; unit: percentage of participants
Arm/Group | Liposomal Bupivacaine | Bupivacaine 0.25%
Number analyzed (Participants) | 20 | 19
percentage of participants | 33.33 | 36.84

7. Secondary Outcome: Sleep Quality
Description: scale of 0-10, 0=horrible, up all night; 10=perfect sleep
Time Frame: Post op Day 1, post op Day 2, post op day 3, post op 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine | Bupivacaine 0.25%
Number analyzed (Participants) | 20 | 19
units on a scale
  Post op Day 1 | 5.06 (3.23) | 3.86 (2.37)
  Post op Day 2 | 6.58 (2.74) | 6 (2.29)
  Post op Day 3 | 6.75 (2.11) | 6.3 (2.46)
  Post Op 1 Week | 7.8 (1.67) | 7.65 (2.49)

ADVERSE EVENTS:
Arm/Group | Liposomal Bupivacaine | Bupivacaine 0.25%
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Bupivacaine (N=20) | Bupivacaine 0.25% (N=19)
ED visit (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes